CLINICAL TRIAL: NCT01976052
Title: Evaluation of Potential Biomarkers for Obstructive Sleep Apnea and the Effect of Positive Pressure Treatment
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Malin Jonsson Fagerlund, MD, PhD, Karolinska University Hospital
Other Study IDs: OSABiomarker
Record Dates: First submitted 2013-10-21; First posted 2013-11-05 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: Biomarkers; Genomics
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Obstructive sleep apnea patients: Patients with obstructive sleep apnea that has not received CPAP treatment
- Matched volunteers with non OSA: Matched volunteers without OSA. Matched in respect to age and BMI
- Matched normal controls with normal BMI: Volunteers that are matched according to age but has a normal BMI

SUMMARY:
Potential biomarkers for obstructive sleep apnea (OSA), and full genomic screening will be evaluated and correlated to the degree of OSA and to effect of CPAP-treatment measured by polygraphy.

DETAILED DESCRIPTION:
This project includes two parts:

* Genomic screening
* Biomarkers

ELIGIBILITY:
OSA-patients with moderate and severe OSA (n=15+15)

1. Adult, 18-75 years of age
2. Moderate (AHI 15-30) or Severe (AHI >30) OSA that are currently untreated and planned for CPAP-treatment
3. Otherwise healthy except for well controlled hypertension since 3 month, Max BP 140/90
4. Non-smokers
5. Not pregnant
6. No medications with antioxidants
7. BMI of <40

Controls (AHI<5) Two groups of controls

1. Matched controls The same age, sex and BMI ± 3 and eventual hypertension. These controls should also fulfill criteria 4-6 above.
2. Healthy controls with normal BMI (19-25) These controls should also fulfill criteria 1., 4-6 above.

Exclusion Criteria:

* If they no not fulfil the inclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: OSA patients will be recruited from an outpatient sleep clinic
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Biomarker | Comparison between 0, 3 and 12 month
  Biomarkers related to inflammation, hypoxia, oxidative stress, redox and the central nervous system will be measured

SECONDARY OUTCOMES:
Genomics | Comparison between 0, 3, 12 month
  Genomic screening by microarray
Apnea hypopnea index | Comparision between 0, 3 and 12 month
  Apnea hypopnea index at 0, 3 and 12 month after treatment with CPAP in the obstructive sleep apnea groups
Exhaled nitric oxide | Comparision at 0, 3 and 12 month
  Measurement of exhaled nitric oxide

CONTACTS AND LOCATIONS:
Overall Officials: Malin Jonsson Fagerlund, MD, PhD, Principal Investigator — Karolinska University Hospital and Karolinska Institutet
Locations (1):
- Department of Anesthesiology, Surgical Sciences and Intensive Care Medicine, Karolinska University Hospital, Solna, Stockholm, Sweden